CLINICAL TRIAL: NCT05501886
Title: Phase 3, Open-Label, Randomized, Study Comparing Gedatolisib Combined With Fulvestrant & With or Without Palbociclib to Standard-of-Care Therapies in Patients With HR-Positive, HER2-Negative Advanced Breast Cancer Previously Treated With a CDK4/6 Inhibitor in Combination w/Non-Steroidal Aromatase Inhibitor Therapy
Brief Title: Gedatolisib Plus Fulvestrant With or Without Palbociclib vs Standard-of-Care for the Treatment of Patients With Advanced or Metastatic HR+/HER2- Breast Cancer (VIKTORIA-1)
Acronym: VIKTORIA-1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Celcuity Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CELC-G-301; 2021-005235-24 (EudraCT Number)
Record Dates: First submitted 2022-08-12; First posted 2022-08-16 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer, Advanced or Metastatic; gedatolisib; HR Positive; ER Positive; HER2 Negative; PIK3CA MT; PI3K
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — gedatolisib; palbociclib; Fulvestrant; Alpelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm A - Patients Lacking PIK3CA Mutations (WT) (Experimental): Gedatolisib + Palbociclib + Fulvestrant
  Interventions: Drug: Gedatolisib; Drug: Palbociclib; Drug: Fulvestrant
- Arm B - Patients Lacking PIK3CA Mutations (WT) (Experimental): Gedatolisib + Fulvestrant
  Interventions: Drug: Gedatolisib; Drug: Fulvestrant
- Arm C - Patients Lacking PIK3CA Mutations (WT) (Active Comparator): Fulvestrant
  Interventions: Drug: Fulvestrant
- Arm D - Patients with PIK3CA Mutation (MT) (Experimental): Gedatolisib + Palbociclib + Fulvestrant
  Interventions: Drug: Gedatolisib; Drug: Palbociclib; Drug: Fulvestrant
- Arm E - Patients with PIK3CA Mutation (MT) (Active Comparator): Alpelisib + Fulvestrant
  Interventions: Drug: Fulvestrant; Drug: Alpelisib
- Arm F - Patients with PIK3CA Mutation (MT) (Experimental): Gedatolisib + Fulvestrant
  Interventions: Drug: Gedatolisib; Drug: Fulvestrant

INTERVENTIONS:
Drug: Gedatolisib — Gedatolisib 180 mg IV given weekly for 3 weeks (Days 1, 8, 15) followed by 1 week off
  Other Names: PF-05212384; PKI-587
  Arms: Arm A - Patients Lacking PIK3CA Mutations (WT); Arm B - Patients Lacking PIK3CA Mutations (WT); Arm D - Patients with PIK3CA Mutation (MT); Arm F - Patients with PIK3CA Mutation (MT)
Drug: Palbociclib — Palbociclib 125 mg PO given daily for 3 weeks (21 days), followed by 1 week off
  Other Names: IBRANCE; PD-0332991
  Arms: Arm A - Patients Lacking PIK3CA Mutations (WT); Arm D - Patients with PIK3CA Mutation (MT)
Drug: Fulvestrant — Fulvestrant 500 mg IM (2 × 5 mL injections) given every 2 weeks during Cycle 1 (Days 1 and 15), then every 4 weeks beginning with Cycle 2 Day 1
  Other Names: Faslodex
Drug: Alpelisib — Alpelisib 300 mg PO (2 × 150 mg tablets) given daily for 4 weeks (28 days)
  Other Names: Piqray; Vijoice; BYL719
  Arms: Arm E - Patients with PIK3CA Mutation (MT)

SUMMARY:
This is a Phase 3, open-label, randomized, clinical trial evaluating the efficacy and safety of gedatolisib plus fulvestrant with or without palbociclib for the treatment of patients with locally advanced or metastatic HR+/HER2- breast cancer following progression on or after CDK4/6 and aromatase inhibitor therapy.

DETAILED DESCRIPTION:
This is a Phase 3, open-label, randomized clinical trial evaluating the efficacy and safety of gedatolisib plus fulvestrant with or without palbociclib for the treatment of patients with advanced (inoperable) or metastatic Hormone Receptor Positive, Human Epidermal Growth Factor Receptor 2 Negative (HR+/HER2-) breast cancer following progression on or after CDK4/6 and aromatase inhibitor therapy. Gedatolisib is an intravenously administered pan-PI3K/mTOR inhibitor. Palbociclib is a CDK4/6 inhibitor. Fulvestrant is a selective estrogen receptor degrader (SERD). Subjects will be assessed for PIK3CA status and then randomized to treatment arms according to their confirmed PIK3CA mutation status.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of metastatic or locally advanced breast cancer Adult females, pre- and/or post-menopausal, and adult males. Pre-menopausal (and peri-menopausal) women can be enrolled if amenable to treatment with an LHRH agonist. Patients are to have commenced concomitant treatment with LHRH agonist prior to or on Cycle 1, Day 1 and must be willing to continue on it for the duration of the study.
2. Negative pregnancy test for women of childbearing potential. Female subjects of childbearing potential must use an effective and/or acceptable contraceptive method from screening until 1 year after the last dose of study treatment
3. Confirmed diagnosis of estrogen receptor positive and/or progesterone receptor positive, as per American Society of Clinical Oncology/College of American Pathologists (ASCO-CAP) guidelines (2020), based on most recent tumor biopsy utilizing an assay consistent with local standards
4. Documented HER2 immunohistochemistry (IHC) negative as per ASCO-CAP 2018 guidance
5. Adequate archival or fresh tumor tissue for the analysis of PIK3CA mutational status
6. Subject must have documentation of radiological disease progression on or after the last prior treatment and also have radiologically evaluable disease (measurable and/or non-measurable) according to RECIST v1.1, per local assessment. Subjects with bone only disease must have lytic or mixed lytic/blastic lesions that can be accurately assessed; bone only blastic lesions with no soft tissue component is not allowed.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
8. Life expectancy of at least 3 months
9. Progressed during or after CDK4/6 inhibitor combination treatment with non-steroidal aromatase inhibitor (AI)
10. Adequate bone marrow, hepatic, renal and coagulation function

Exclusion Criteria:

1. History of malignancies other than adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for ≥3 years
2. Prior treatment with a phosphoinositide 3-kinase (PI3K) inhibitor, a protein kinase B (Akt) inhibitor, or a mechanistic target of rapamycin (mTOR) inhibitor
3. Prior treatment with chemotherapy and antibody drug conjugates for advanced disease is not permitted (prior adjuvant or neoadjuvant chemotherapy is permitted)
4. More than 2 lines of prior endocrine therapy treatment
5. Bone only disease that is only blastic with no soft tissue component
6. Subjects with type 1 diabetes or uncontrolled type 2 diabetes
7. Known and untreated, or active, brain or leptomeningeal metastases

   a. Subjects with previously treated central nervous system (CNS) metastases may be enrolled in the study if they meet the following criteria: do not require supportive therapy with steroids; do not have seizures and do not exhibit uncontrolled neurological symptoms; stable disease confirmed by radiographic assessment within at least 4 weeks prior to enrollment
8. Patients with advanced, symptomatic, visceral spread that are at risk of life-threatening complication in the short-term
9. History of clinically significant cardiovascular abnormalities such as: Congestive heart failure (New York Heart Association (NYHA) classification ≥ II within 6 months of study entry

   1. Myocardial infarction within 12 months of study entry
   2. History of any uncontrolled (or untreated) clinically significant cardiac arrhythmias, (e.g., ventricular tachycardia), complete left bundle branch block, high grade AV block (e.g., bifascicular block, Mobitz type II and third degree AV block), supraventricular, nodal arrhythmias, or conduction abnormality in the previous 12 months
   3. Uncontrolled hypertension defined by systolic blood pressure (SBP) ≥160 mmHg and/or diastolic blood pressure (DBP) ≥100 mmHg, with or without antihypertensive medication (initiation or adjustment of antihypertensive medication[s] is allowed prior to screening)
   4. Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:

      * i. Risk factors for Torsades de Pointes (TdP) including uncorrected hypokalemia or hypomagnesemia, or history of clinically significant/symptomatic bradycardia
      * ii. On screening, inability to determine the corrected QT interval using Fridericia's formula (QTcF) on the ECG (i.e., unreadable or not interpretable) or QTcF >480 msec (determined by mean of triplicate ECGs at screening)
10. Known hypersensitivity to the study drugs or their components
11. Pregnant or breast-feeding women
12. Concurrent participation in another interventional clinical trial

    1. Subjects must agree not to participate in another clinical trial (other than observational) at any time during participation in VIKTORIA-1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 701 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) in Patients with PIK3CA WT and PIK3CA MT Breast Cancer | Approximately 48 months
  PFS is defined as the time from randomization to death or the first documented progression, whichever occurs first, confirmed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria, as determined based on blinded independent central review (BICR)

SECONDARY OUTCOMES:
Overall Survival (OS) in Patients with PIK3CA WT and PIK3CA MT Breast Cancer | From date of randomization to the date of death due to any cause, up to approximately 48 months
  OS is defined as the length of time from randomization until the date of death from any cause method, where PFS is defined as the time from randomization to death or the first documented progression, whichever occurs first, confirmed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria, as determined based on blinded independent central review (BICR)
Overall Response Rate (ORR) in Patients with PIK3CA WT and PIK3CA MT Breast Cancer | Up to approximately 48 months
  Percentage of subjects who achieved an objective response according to RECIST v1.1 criteria (complete response [CR] or partial response [PR]) as assessed by BICR)
Duration of Response (DOR) in Patients with PIK3CA WT and PIK3CA MT Breast Cancer | Up to approximately 48 months
  Time from the assessment of initial response (PR or better) to death or first documented disease progression as assessed by BICR, whichever occurs first
Time to Response (TTR) in Patients with PIK3CA WT and PIK3CA MT Breast Cancer | Up to approximately 48 months
  Time form randomization to the first assessment of PR or better as assessed by BICR, whichever comes first
Clinical Benefit Rate (CBR) in Patients with PIK3CA WT and PIK3CA MT Breast Cancer | Up to approximately 48 months
  Percentage of subjects with CR, PR, or stable disease (SD) >24 weeks as assessed by BICR
Quality of Life (QOL)Functional Assessment of Cancer Therapy - Breast Trial Outcome Index (FACT-B TOI) Questions in Patients with PIK3CA WT and PIK3CA MT Breast Cancer | From baseline to 30 Day Safety Follow-up
  The FACT-B TOI is an abbreviated (24-item) version of the full FACT-B which focuses only on the patient's Physical Well-being (PWB), Functional Well-being (FWB), and Breast Cancer Subscale (BCS) components using a 5-level scale, (Not at all, A little bit, Some-what, Quite a bit, Very much).
Quality of Life (QOL) NCCN-FACT Breast Symptom Index -16 (NFBSI-16) in Patients with PIK3CA WT and PIK3CA MT Breast Cancer | From baseline to 30 Day Safety Follow-up
  NCCN-FACT is derived from the FACT-B and only 4 additional items will be administered to enable optional scoring of the NFBSI subscales and total score using a 5-level scale (Not at all, A little bit, Some-what, Quite a bit, Very much).
Patient-Reported Outcomes in Patients with PIK3CA WT and PIK3CA MT Breast Cancer | From baseline to 30 Day Safety Follow-up
  Patient-Reported Outcomes Measurement Information System (PROMIS®) Short Form v2.0 - Physical Function 8c using a 5-level scale (Without any difficulty, With a little difficulty, With some difficulty, With much difficulty, Unable to do)
EuroQol 5 in Patients with PIK3CA WT and PIK3CA MT Breast Cancer | From baseline to 30 Day Safety Follow-up
  EuroQol 5 Dimension 5 Level (EQ-5D-5L) - This is a 5 question, self-administered visual analog scale (VAS) where patients use 0 (worst health) to 100 (best health) to indicate how they view their health.
Adverse Events | Up to approximately 48 months
  Safety and tolerability will be evaluated by review of type, incidence, severity (as graded by the National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] v5.0), seriousness, and relationship to study medications of adverse events (AEs) and any laboratory abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Nadene Zack, Study Director — Celcuity Inc
Locations (235):
- United States (71):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Oncology (US Oncology/McKesson) - Goodyear, Goodyear, Arizona
  - St. Bernards Medical Center, Jonesboro, Arkansas
  - CARTI Cancer Center, Little Rock, Arkansas
  - Pacific Cancer Medical Center Inc, Anaheim, California
  - Kaiser Permanente South Bay Medical Center, Harbor City, California
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - Pacific Cancer Care, Monterey, California
  - University of California, Irvine Medical Center, Orange, California
  - Ventura County Hematology Oncology Specialists, Oxnard, California
  - Redlands Hematology Oncology, Redlands, California
  - UCLA Hematology/Oncology-Santa Monica, Santa Monica, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - PIH Health Hospital Whittier, Whittier, California
  - Yale Cancer Center - New Haven, New Haven, Connecticut
  - South Broward Hospital District d/b/a Memorial Healthcare System, Hollywood, Florida
  - Cancer Specialists of North Florida - Jacksonville, Jacksonville, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Bond & Steele Clinic, P.A. d/b/a Bond Clinic, P.A., Winter Haven, Florida
  - John D. Archbold Memorial Hospital, Thomasville, Georgia
  - Illinois Cancer Specialists - Arlington Heights, Arlington Heights, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - University of Kansas Cancer Center, Westwood, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Mercy Health - Paducah, Paducah, Kentucky
  - American Oncology Partners of Maryland, PA, Bethesda, Maryland
  - Maryland Oncology Hematology, P.A. - Rockville, Rockville, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Nebraska Hematology - Oncology, P.C., Lincoln, Nebraska
  - Oncology Hematology West PC dba Nebraska Cancer Specialists, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - New York Oncology Hematology, P.C. - Albany, Albany, New York
  - Queens Hospital Cancer Center, Jamaica, New York
  - Coleman, Pasmantier & Decter, MDs, New York, New York
  - Weill Cornell Medicine/New York-Presbyterian Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Hematology/Oncology Associates of Central New York, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - White Plains Hospital, White Plains, New York
  - Cone Health Cancer Center at Alamance Regional, Hematology/Oncology, Greensboro, North Carolina
  - Southeast Regional Cancer Center, Lumberton, North Carolina
  - Sanford Health- Fargo, Fargo, North Dakota
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Oregon Oncology Specialists, Salem, Oregon
  - Northwest Cancer Specialists, PC - Tigard, Tigard, Oregon
  - Consultants In Medical Oncology and Hematology, P.C., Broomall, Pennsylvania
  - Alliance Cancer Specialists PC, Horsham, Pennsylvania
  - Cancer Care Associates of York, York, Pennsylvania
  - Sanford Gynecologic Oncology Clinic, Sioux Falls, South Dakota
  - Texas Oncology - Austin, Austin, Texas
  - Texas Oncology P.A. - Dallas, Dallas, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - William Beaumont Army Medical Center, El Paso, Texas
  - Oncology Consultants, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Brooke Army Medical Center, Houston, Texas
  - Texas Oncology - McKinney, McKinney, Texas
  - Texas Oncology - Gulf Coast, Sugar Land, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Fort Belvoir Community Hospital, Fort Belvoir, Virginia
  - Bon Secours St. Francis Medical Oncology Center, Midlothian, Virginia
  - Virginia Oncology Associates - Newport News, Newport News, Virginia
  - VCU Massey Cancer Center, Richmond, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care - Roanoke, Roanoke, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Northwest Medical Specialties, PLLC - Tacoma, Tacoma, Washington
- Argentina (13):
  - CENIT Foundation, Buenos Aires
  - Alexander Fleming Institute, Buenos Aires
  - Buenos Aires British Hospital, Buenos Aires
  - Center for Medical Education and Clinical Research (CEMIC), Buenos Aires
  - Fleischer Medical Center, Buenos Aires
  - Medical Center Austral, Buenos Aires
  - Pergamino Clinic, Buenos Aires
  - Cordoba Oncology Institute (IONC), Córdoba
  - Center of Nuclear and Molecular Medicine of Entre Rios (CEMENER), Paraná
  - CEDIT Diagnostic and treatment center, Salta
  - CER San Juan, San Juan
  - 9 of July Sanatorium, San Miguel de Tucumán
  - Rosario's Oncology Institute and Medical Specialities (IOR), Santa Fe
- Australia (8):
  - Adelaide Oncology & Haematology, Adelaide
  - St Vincent's Hospital (Melbourne) Ltd, Fitzroy
  - Peninsula & South Eastern Hematology and Oncology Group (PSEHOG), Frankston
  - Hollywood Private Hospital, Breast Cancer Research Centre, Nedlands
  - Mater Hospital Brisbane, Mater Cancer Care Centre, South Brisbane
  - Icon Cancer Centre- Southport, Southport
  - Sydney Adventist Hospital, Wahroonga
  - The Queen Elizabeth Hospital, Woodville
- Austria (8):
  - University Hospital Graz, Department of Gynecology and Obstetrics, Graz
  - University Hospital Innsbruck - Tyrolean Hospital, Department of Gynaecology and Obstetrics, Innsbruck
  - Order Hospital Linz Ltd. - Hospital of Sisters of Mercy, Department of Internal Medicine I, Linz
  - Salzburg Regional Hospital, Department of Internal Medicine III, Salzburg
  - University Hospital St. Poelten, Department of Internal Medicine I, Sankt Pölten
  - Hospital Hietzing, Department of Gynecology, Vienna
  - Medical University Vienna, Department of Gynecology and Obstetrics, Vienna
  - Hospital Wels-Grieskirchen, Internal Medicine Department IV, Wels
- Belgium (9):
  - Saint Luc University Hospital, Brussels
  - Charleroi Grand Hospital (GHDC), Charleroi
  - University Hospital Antwerp (UZA), Edegem
  - AZ Groeninge, Kortrijk
  - University Hospitals Leuven, Campus Gasthuisberg, Leuven
  - Citadelle Regional Hospital Center, Liège
  - VITAZ, Sint-Niklaas
  - Centre Hospitalier Peltzer-la-Tourelle, Verviers
  - UCL Mont-Godinne University Hospitals, Yvoir
- Brazil (9):
  - Oncology Treatment Center, Belém, Pará
  - Catarina Clinical Research, Itajaí, Santa Catarina
  - Pronutrir, Fortaleza
  - ONCOSITE - Clinical Research Center in Oncology, Ijuí
  - Juiz de Fora Eurolatino Research Center, Minas Gerais
  - Bahia Oncology Center, Salvador
  - Portuguese Sao Paulo Charity / Sao Jose Hospital, São Paulo
  - D'OR Institute, São Paulo
  - Hospital A.C.Camargo, São Paulo
- Bulgaria (5):
  - Multiprofile Hospital for Active Treatment - Uni Hospital, Panagyurishte, Panagyurishte
  - MHAT for Women's Health "Nadezhda", Sofia
  - Multiprofile Hospital for Active Treatment "Serdika", Sofia, Sofia
  - Specialized Hospital for Active Treatment in Oncology, Clinic of Medicial Oncology (Chemotherapy), Sofia
  - University Multiprofile Hospital for Active Treatment "Sveta Marina", Varna
- Canada (5):
  - BC Cancer - Vancouver, Medical Oncology, Vancouver, British Columbia
  - Walker Family Cancer Center, St. Catharines, Ontario
  - CIUSSS du Saguenay Lac St-Jean, Chicoutimi, Quebec
  - Hospital Notre-Dame, Montreal, Quebec
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
- Czechia (4):
  - University Hospital Olomouc, Clinic of Oncology, Olomouc
  - Thomayer University Hospital, Clinic of Oncology, Prague
  - University Hospital Bulovka, Institute of Radiation Oncology, Prague
  - University Hospital Motol, Clinic of Oncology, Prague
- France (7):
  - Bergonie Institute, Bordeaux
  - Francois Baclesse Center, Caen
  - La Roche-sur-Yon Hospital, La Roche-sur-Yon
  - CHU La Timone - La Timone Children's Hospital, Marseille
  - University Hospital Center of Poitiers, Poitiers
  - Saint Anne Clinic, Strasbourg
  - Gustave Roussy, Villejuif
- Germany (8):
  - Hospital Bayreuth, Bayreuth
  - Vivantes Hospital Am Urban, Berlin
  - Hospital Suedstadt Rostock, Dorf Mecklenburg
  - Private Practice with Focus on Oncology, Lübeck
  - University Hospital Johannes Gutenberg - University of Mainz, Mainz
  - University Hospital Muenster, Münster
  - Caritas Klinikum, Saarbrücken
  - Helios Clinic Wuppertal, Wuppertal
- Greece (10):
  - Metropolitan General Hospital, Athens
  - Alexandra General Hospital, Athens
  - University General Hospital of Ioannina, Ioannina
  - University General Hospital of Larissa, Larissa
  - IASO Thessaly SA, Larissa
  - Metropolitan Hospital, Piraeus
  - Bioclinic Thessalonikis S.A., Thessaloniki
  - European Interbalkan Medical Center of Thessaloniki, Thessaloniki
  - EUROMEDICA General Clinic of Thessaloniki, Thessaloniki
  - Theageneio Anticancer Hospital of Thessaloniki, Thessaloniki
- Hungary (3):
  - University of Debrecen Clinical Center, Institute of Oncology, Debrecen
  - Bacs-Kiskun County Hospital, Center for Oncoradiology, Kecskemét
  - Szabolcs-Szatmar-Bereg County Hospitals and University Teaching Hospital, Department of Oncology, Nyíregyháza
- India (6):
  - Shri Ram Cancer Centre, Mahatma Gandhi Medical College & Hospital, Jaipur, Rajasthan
  - HCG Cancer Centre, Bangalore
  - Postgraduate Institute of Medical Education and Research (PGIMER), Chandigarh
  - Tata Medical Center, Kolkata
  - Tata Memorial Hospital, Navi Mumbai
  - Christian Medical College, Department of Medical Oncology, Vellore
- Italy (8):
  - European Institute of Oncology (IEO), IRCCS, Milan
  - University Polyclinic Hospital of Modena, Modena
  - Local Healthcare Company of Monza (ASST Monza), Monza
  - University Hospital of Parma, Parma
  - New Hospital of Prato (NOP), Prato
  - University Hospital Campus Bio-Medico, Rome
  - University Polyclinic Foundation "Agostino Gemelli" - IRCCS, Rome
  - Santa Maria della Misericordia University Hospital of Udine, Udine
- Mexico (9):
  - Clinical Research Center Chapultepec Mexico City, Mexico City
  - CRYPTEX, Mexico City
  - ProcliniQ Clinical Research, Mexico City
  - Filios High Medicine, Monterrey
  - Administrative Society of Health Services, SC, Morelia
  - Avix Clinical Research, Nuevo León
  - Zambrano Hellion Medical Center, Nuevo León
  - Inbiomedyc, Querétaro
  - ONCOR Life Medical Center, Saltillo
- Poland (10):
  - Prof. Franciszek Lukaszczyk Oncology Center in Bydgoszcz, Chemotherapy Outpatient Clinic, Bydgoszcz
  - Medical Clinic "Komed", Konin
  - Maria Sklodowska-Curie Institute of Oncology, Branch in Krakow, Krakow
  - Polish Mother's Memorial Hospital-Research Institute, Lodz
  - Independent Public Healthcare Facility Prof. Tadeusz Koszarowski Opole Oncology Center in Opole, Clinical Oncology Department and Day Hospitalization Unit, Opole
  - St. John Paul 2nd Mazovian Provincial Hospital in Siedlce Limited Liability Company, Siedlce Oncology Centre, Siedlce
  - West Pomeranian Oncology Center, Szczecin
  - LUX MED Oncology LLC, Szamocka Hospital, Department of Clinical Oncology/Chemotherapy, Warsaw
  - Maria Sklodowska-Curie - National Research Institute of Oncology, Warsaw
  - Provincial Specialist Hospital in Wroclaw, Department of Chemotherapy, Wroclaw
- Romania (8):
  - S.C. Oncopremium-Team SRL, Baia Mare
  - Prof. Dr. Alexandru Trestioreanu Institute of Oncology, Bucharest
  - "Prof. Dr. Ion Chiricuta" Institute of Oncology, Radiotherapy Department I, Cluj-Napoca
  - Prof. Dr. Ion Chiricuta Institute of Oncology, Cluj-Napoca
  - Onco Clinic Consult S.A., Craiova
  - Oncology Center "Sf. Nectarie", Craiova
  - S.C. Radiotherapy Center Cluj SRL, Department of Medical Oncology, Floreşti
  - S.C. Topmed Medical Center SRL, Târgu Mureş
- Singapore (5):
  - Curie Oncology, Singapore
  - ICON SOC Farrer Park Medical Clinic, Singapore
  - OncoCare Cancer Centre, Singapore
  - Raffles Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Korea (6):
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Soeul
  - Korea University Anam Hospital, Soeul
  - Samsung Medical Center, Soeul
  - Severance Hospital, Yonsei University Health System, Soeul
  - Ulsan University Hospital, Ulsan
- Spain (8):
  - University Hospital Ramon y Cajal, Madrid, Madrid
  - Infanta Cristina Hospital, Badajoz
  - Catalan Institute of Oncology, Hospital Duran i Reynals, Barcelona
  - Caceres Hospital Complex - San Pedro de Alcantara General Hospital, Cáceres
  - Hospital Ruber Internacional, Madrid
  - University Hospital Foundation Jimenez Diaz, Madrid
  - University Clinical Hospital Virgen de la Arrixaca, Department of Oncology, Murcia
  - University Hospital Complex of Santiago (CHUS), Department of Oncology, Santiago de Compostela
- Taiwan (8):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taipei Medical University - Shuang Ho Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - National Taiwan University Hospital - Yunlin Branch (Huwei District), Yuanlin
- United Kingdom (7):
  - Royal United Hospital, Department of Oncology/Hematology, Bath
  - Velindre Cancer Centre, Cardiff
  - Guy's Hospital, London
  - Royal Marsden Hospital - London, Department of Medical Oncology, London
  - The Christie NHS Foundation Trust, Manchester
  - Nottingham City Hospital, Nottingham
  - Royal Marsden Hospital - Sutton, Sutton